CLINICAL TRIAL: NCT04846946
Title: Conducting the Preparation Phase of a Multiphase Optimization Strategy (MOST) to Develop a Modular HIV Prevention and PrEP Intervention for Sexual and Gender Minority Adolescents and Parents: "Hey, Friend"
Brief Title: HIV Prevention and PrEP Intervention for SGM Adolescents and Parents: "Hey, Friend"
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Opted to not conduct this study; revised to a more condensed study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Henna Budhwani, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MISP #60819
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: HIV Infections
Keywords: HIV; PrEP
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: In Aim 3 of our study, our goal is to complete the MOST preparation phase wherein we collect acceptability, feasibility, and some effectiveness data on each module prior to combining them to test the effects of the full intervention package.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Time attention control condition.
- Intervention, Module 1 - Knowledge (Experimental): 20-minute module that aims to improve HIV prevention knowledge.
  Interventions: Behavioral: Hey, Friend
- Intervention, Module 1 - Stigma (Experimental): 20-minute module that aims to reduce SGM- and HIV- related stigma.
  Interventions: Behavioral: Hey, Friend
- Intervention, Module 1 - Prevention (Experimental): 20-minute module that aims to promote HIV prevention strategies including testing and PrEP.
  Interventions: Behavioral: Hey, Friend

INTERVENTIONS:
Behavioral: Hey, Friend — Intervention in development. However, we will use intervention mapping and the designing for dissemination approach, informed by self-reported qualitative data, to develop the "Hey, Friend" modules. The mHealth intervention will include three modules that include multiple sub-topics (e.g., What is HIV?; How do I protect myself from HIV?; What is PrEP?, etc.), deliver culturally appropriate counseling content in community settings, juvenile court system, clinics, and schools; will include Motivational Interviewing components that are effective in evoking behavior change while being acceptable to adolescents and parents, and will include ongoing support through a text reminder to maximize the likelihood of initiating HIV prevention through testing and PrEP.
  Arms: Intervention, Module 1 - Knowledge; Intervention, Module 1 - Prevention; Intervention, Module 1 - Stigma

SUMMARY:
In this 24-month pilot study, we will conduct the preparation phase of a multiphase optimization strategy (MOST) to develop a culturally appropriate (for Deep South contexts, to be adolescent friendly, and to be acceptable to parents or guardians) modular HIV prevention mHealth intervention, targeting behavior change related to HIV testing, HIV prevention knowledge, and pre-exposure prophylaxis (PrEP) uptake for sexual and gender minority (SGM) adolescents, that can be seamlessly integrated into the existing school and community environments across the Deep South.

DETAILED DESCRIPTION:
In this 24-month pilot study, we will conduct the preparation phase of a multiphase optimization strategy (MOST) to develop a culturally appropriate (for Deep South contexts, to be adolescent friendly, and to be acceptable to parents or guardians) modular HIV prevention mHealth intervention, targeting behavior change related to HIV testing, HIV prevention knowledge, and pre-exposure prophylaxis (PrEP) uptake for sexual and gender minority (SGM) adolescents, that can be seamlessly integrated into the existing school and community environments across the Deep South. To do so, in Aim 1, we will assess stakeholders' knowledge, sentiments, and beliefs related to HIV risk, HIV stigma, and HIV prevention including preferences related to modality of PrEP and PrEP acceptability. Then, in Aim 2, we will use Aim 1 data, applying the 4-step intervention mapping framework, to inform the development of intervention modules targeting 14-18 year old SGM adolescents (rationale for this age range presented later in this proposal). We will also, develop corollary modules for parents or guardians. After intervention modules have been finalized, in Aim 3, we will conduct a 4-arm randomization to assess each module's acceptability, feasibility, and clinical signal of effectiveness as compared to a time-attention control.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 14-18
* Parental or guardian consent
* SGM identity
* English speaking

Exclusion Criteria:

* Does not fit the inclusion criteria

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
HIV Knowledge | Year 2
  HIV Knowledge Questionnaire (HIV-K-Q), Scored 0-18 with 18 indicating thorough HIV knowledge and 0 indicating no HIV knowledge
SGM Related Stigma | Year 2
  Perceived Racism Scale (PRS). Scores for the PRS frequency of exposure scale can range from 0 to 301; higher scores indicate more frequent perceptions of exposure to racism.
HIV Testing Behaviors | Year 2
  Binary Yes or No to Accept an HIV Test after Module

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham (UAB), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
We do not intend to share IPD.